CLINICAL TRIAL: NCT00410020
Title: Secondary Prevention of Atrial Fibrillation With an Alpha-Linolenic Enriched Diet : a Randomized Study
Brief Title: Arrhythmia Prevention With an Alpha-Linolenic Enriched Diet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University Hospital, Bordeaux (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DGS 990321; 99-04 (CPPRB BORDEAUX B)
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2006-12-12 (Estimated); Status verified 2006-12

CONDITIONS: Atrial Fibrillation; Diet Therapy
Keywords: alpha linolenic acid; atrial fibrillation; omega 3 fatty acids; diet; rapeseed oil; canola oil; cardiovascular diseases
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases

INTERVENTIONS:
Behavioral: Alpha-linolenic enriched diet

SUMMARY:
An alpha linolenic acid (ALA) rich diet in the Lyon Diet Heart Study reduced sudden cardiac deaths possibly by reducing cardiac arrhythmias and ventricular fibrillation (Lancet 1994).

Since then, there has been a growing interest in ALA, ω-3 fatty acid family precursor, as a cardioprotective nutrient. Much of the interest has focused on the potential antiarrhythmic effect of longer chain ω-3 fatty acids, DHA and EPA, derived from fish.

We therefore concluded it important to test wether vegetable source ω-3 also had antiarrhythmic effects, as shown in animals by Leaf and McLennan, since this might also explain the beneficial effects seen on cardiovascular mortality in the Lyon Diet Heart Study.

DETAILED DESCRIPTION:
Objective: To determine the effect of an ALA rich diet in reducing recurrence of atrial fibrillation as a further example of a cardiac arrhythmia.

Design: Randomized parallel design efficacy study.

Setting: Three university hospital centers in the Bordeaux region, France.

Patients: 98 patients randomized immediately after successful atrial fibrillation electrical cardioversion.

Intervention: A canola margarine and oil, versus a conventional diet (control), with a one year follow-up.

Main outcome measure: Length of time to first recurrence of atrial fibrillation.

Significance: If ALA is antiarrhythmic, this action may explain its cardioprotective effect in clinical trials and cohort studies.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in one of the three centers in the Bordeaux region
* clinical diagnosis of atrial fibrillation
* who subsequently underwent successful electrical cardioversion

Exclusion Criteria:

* unable to receive electrical cardioversion
* already enrolled in another trial
* unable or unwilling to comply with the diet recommendations (experimental or control) or follow-up requirements
* clinically significant cardiac disease, advanced heart failure, cardiac cachexia
* thyroid disease, treated or untreated,
* clinically significant hepatic or renal disease
* history of malignant disease
* alcohol abuse
* taking ALA rich foods or recording intakes of ALA >2g/d on the control diet or reporting using <1g/d on the ALA diet was considered a major deviation from the protocol

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 1999-06; Study Completion 2003-06

PRIMARY OUTCOMES:
Rate of recurrence on periods
Length of time to first recurrence of atrial fibrillation

SECONDARY OUTCOMES:
subgroup analysis (high blood pressure, non persistent atrial fibrillation)
comparison between late and early recurrence (before or after 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Broustet, MD, PhD, Principal Investigator — Universitary Hospital Haut-Lévêque Bordeaux France; Serge C Renaud, VMD, PhD, Study Chair — Bordeaux2 University; Dominique Lanzmann-Petithory, MD, PhD, Study Director — Bordeaux2 University - Paris AP Hospitals
Locations (3):
- France (3):
  - Girac Hospital, Angoulême
  - Hôpital du Haut-Lévêque, Bordeaux
  - Robert Boulin Hospital, Libourne

REFERENCES:
- [Background] de Lorgeril M, Renaud S, Mamelle N, Salen P, Martin JL, Monjaud I, Guidollet J, Touboul P, Delaye J. Mediterranean alpha-linolenic acid-rich diet in secondary prevention of coronary heart disease. Lancet. 1994 Jun 11;343(8911):1454-9. doi: 10.1016/s0140-6736(94)92580-1. PMID 7911176
- [Background] Renaud S, de Lorgeril M, Delaye J, Guidollet J, Jacquard F, Mamelle N, Martin JL, Monjaud I, Salen P, Toubol P. Cretan Mediterranean diet for prevention of coronary heart disease. Am J Clin Nutr. 1995 Jun;61(6 Suppl):1360S-1367S. doi: 10.1093/ajcn/61.6.1360S. PMID 7754988
- [Background] Renaud S, Nordoy A. "Small is beautiful": alpha-linolenic acid and eicosapentaenoic acid in man. Lancet. 1983 May 21;1(8334):1169. doi: 10.1016/s0140-6736(83)92902-1. No abstract available. PMID 6133188
- [Background] Lanzmann-Petithory D, Pueyo S, Renaud S. Primary prevention of cardiovascular diseases by alpha-linolenic acid. Am J Clin Nutr. 2002 Dec;76(6):1456; author reply 1456-7. doi: 10.1093/ajcn/76.6.1456. No abstract available. PMID 12450919
- [Background] Renaud SC, Lanzmann-Petithory D. alpha-linolenic acid in the prevention of cardiovascular diseases. World Rev Nutr Diet. 2001;88:79-85. doi: 10.1159/000059769. No abstract available. PMID 11935975
- [Background] Renaud SC, Lanzmann-Petithory D. The beneficial effect of alpha-linolenic acid in coronary artery disease is not questionable. Am J Clin Nutr. 2002 Oct;76(4):903-4; author reply 904-6. doi: 10.1093/ajcn/76.4.903. No abstract available. PMID 12324307
- [Background] Singh RB, Dubnov G, Niaz MA, Ghosh S, Singh R, Rastogi SS, Manor O, Pella D, Berry EM. Effect of an Indo-Mediterranean diet on progression of coronary artery disease in high risk patients (Indo-Mediterranean Diet Heart Study): a randomised single-blind trial. Lancet. 2002 Nov 9;360(9344):1455-61. doi: 10.1016/S0140-6736(02)11472-3. PMID 12433513
- [Background] Lanzmann-Petithory D. Alpha-linolenic acid and cardiovascular diseases. J Nutr Health Aging. 2001;5(3):179-83. PMID 11458289
- [Background] Kang JX, Leaf A. Protective effects of free polyunsaturated fatty acids on arrhythmias induced by lysophosphatidylcholine or palmitoylcarnitine in neonatal rat cardiac myocytes. Eur J Pharmacol. 1996 Feb 15;297(1-2):97-106. doi: 10.1016/0014-2999(95)00701-6. PMID 8851173
- [Background] McLennan PL, Dallimore JA. Dietary canola oil modifies myocardial fatty acids and inhibits cardiac arrhythmias in rats. J Nutr. 1995 Apr;125(4):1003-9. doi: 10.1093/jn/125.4.1003. PMID 7722678